CLINICAL TRIAL: NCT07171528
Title: Secondary Cytoreductive Surgery After Chemotherapy for Recurrent Epithelial Ovarian Cancer: A Phase II Randomized Controlled Trial
Brief Title: Secondary Cytoreductive Surgery After Chemotherapy for Recurrent Epithelial Ovarian Cancer
Acronym: KOV-02S
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, MD, PhD, Principal Researcher, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2025-0092
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Recurrent ovarian cancer; Epithelial Ovarian Cancer; platinum sensitive recurrent ovarian cancer; secondarycytoreductive surgery
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Participants are aware of their group assignment in this open-label randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Secondary Cytoreductive Surgery (No Intervention): * Secondary cytoreductive surgery in this study will be performed in patients who have undergone 3 cycles of chemotherapy and shown a response (Complete response, partial response, or stable disease).
  * The chemotherapy regimen used before and after the intervention will be the same. Chemotherapy for patients with progressive ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that recurs at least 6 months after platinum-based chemotherapy will be used.
  * Both the CRS group and the control group will receive adjuvant chemotherapy for 3-6 cycles after enrollment.
  * The following chemotherapy regimens are allowed and correspond to the standard treatments for platinum-sensitive recurrent ovarian cancer:
    * Carboplatin/Paclitaxel ± Bevacizumab
    * Carboplatin/Liposomal Doxorubicin ± Bevacizumab
    * Carboplatin/Gemcitabine ± Bevacizumab
    * Carboplatin/Topotecan
    * Cisplatin/Topotecan
    * Carboplatin/Docetaxel
    * Cisplatin/Docetaxel
- Secondary Cytoreductive Surgery (Experimental): Surgery will only be performed in patients assigned to the experimental arm of the study.
  The goal of secondary cytoreductive surgery is to achieve complete tumor reduction by removing all visible residual tumors (Complete cytoreduction with no macroscopic residual disease), and this effort should be the top priority.
  Interventions: Procedure: Secondary Cytoreductive Surgery

INTERVENTIONS:
Procedure: Secondary Cytoreductive Surgery — Surgery will only be performed in patients assigned to the experimental arm of the study.
  The goal of secondary cytoreductive surgery is to achieve complete tumor reduction by removing all visible residual tumors (Complete cytoreduction with no macroscopic residual disease), and this effort should be the top priority.
  Arms: Secondary Cytoreductive Surgery

SUMMARY:
To compare outcomes between the CRS group and the control group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy

DETAILED DESCRIPTION:
[Primary Objective] To compare the progression-free survival (PFS) between the CRS group and the control group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.

[Secondary Objectives]

1. To compare the overall survival (OS) and cancer-specific survival (CSS) between the CRS group and the control group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.
2. To evaluate the adverse events between the CRS group and the control group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.
3. To assess the quality of life (QoL) between the CRS group and the control group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.
4. To investigate the prognostic role of the CA-125 KELIM model in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.
5. To perform a cost-effectiveness analysis of the CRS group in patients with recurrent epithelial ovarian cancer who have undergone chemotherapy.

ELIGIBILITY:
[Inclusion Criteria]

1. Patients with histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
2. Patients with recurrent ovarian cancer who have received platinum-based chemotherapy (3 or 4 cycles) and were deemed unsuitable for secondary cytoreductive surgery due to a negative AGO score according to the DESKTOP-III trial.
3. Patients with recurrent ovarian cancer who have responded to chemotherapy (Complete Response, Partial Response, or Stable Disease).
4. The patient's disease must have recurred after platinum-based therapy, and be defined as platinum-sensitive, meaning progression occurred more than 6 months (180 days) after the last administration of platinum-based therapy.
5. Patients aged 19 years or older at the time of providing informed written consent.
6. Patients with an ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2 within 28 days prior to clinical trial allocation.
7. Women who are medically unable to conceive or, if of childbearing potential, must agree to follow contraception guidelines during the treatment period.
8. The participant (or their legally authorized representative) must provide informed written consent regarding the trial.
9. The participant may consent to the secondary use of clinical information for future biomedical research. However, refusal to share clinical information for future research does not affect participation in the main trial.
10. The participant must have adequate organ function as defined in the table below. Specimens must be collected within 28 days.

1) Adequate bone marrow function defined as

* White Blood Cell (WBC)≥ 2,500/㎕
* Platelet (PLT)≥ 100,000/㎕
* Hemoglobin (H)≥ 8 g/dl (after correction in cases of simple iron-deficiency anemia) 2) Adequate renal function defined as
* Creatinine or Creatinine Clearance (Cr or CrCl) or Glomerular filtration rate (GFR) (GFR can also be used instead of Cr or CrCl)

  * Creatinine ≤ 1.5 mg/dL or within 1.5 times the upper limit of normal (ULN)
  * CrCl ≥ 30 mL/min or GFR-EPI ≥ 30 mL/min/1.73m² 3) Adequate liver function defined as
* Total Bilirubin≤ 1.5 x ULN
* AST (SGOT) and ALT (SGPT)≤ 2.5 x ULN (for patients with liver metastasis, ≤ 5.0 x ULN) 4) No Significant dysfunction in Heart, Lungs, etc.

  * No abnormalities in preoperative pulmonary function tests, electrocardiograms (ECG), or chest X-rays.
  * For patients with a history of cardiac or pulmonary diseases, a collaborative evaluation with cardiology or pulmonology must confirm that surgery is feasible.

ALT(SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase) AST(SGOT) = aspartate aminotransferase (serum glutamic oxaloacetic transaminase) GFR = glomerular filtration rate; ULN = upper limit of normal

[Exclusion Criteria]

1. Patients with non-epithelial ovarian cancer or borderline ovarian tumors.
2. Patients with recurrent ovarian cancer who are not suitable for platinum-based chemotherapy.
3. Patients over 80 years of age.
4. Patients with a clinically assessed life expectancy of less than 3 months.
5. Patients deemed unsuitable for secondary cytoreductive surgery due to clinical findings (e.g., severe adhesions, bowel obstruction, fistula, perforation, or other conditions making surgery infeasible).
6. Patients with inadequate, cardiac, pulmonary, hepatic, renal, or bone marrow function for surgery.
7. Patients with uncontrolled active infections.
8. Patients diagnosed with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML), or those exhibiting features suggestive of MDS/AML.
9. Patients whose primary disease is an extra-abdominal condition that is expected to be a major cause of morbidity or mortality.
10. Patients with active central nervous system metastasis or carcinomatous meningitis. Patients with a history of brain metastasis must be radiologically stable.
11. Patients with infections requiring systemic treatment (parenteral administration of antibiotics for bacterial, antifungal, or antivirals).
12. Patients with uncontrolled active tuberculosis (TB) within one month before treatment initiation.
13. Patients with psychiatric disorders that may interfere with their ability to comply with the trial, including those diagnosed with mental illness or substance abuse disorders.
14. Female patients who have not undergone a hysterectomy and have a positive urine pregnancy test within 14 days prior to study allocation. For women of childbearing potential, even if the screening urine pregnancy test is negative, additional pregnancy tests may be conducted at the discretion of the investigator at the time of surgery or chemotherapy initiation Pregnancy tests are not required for women who have undergone hysterectomy or are otherwise confirmed to be infertile.
15. Patients who are currently breastfeeding.
16. Patients with a history of allogeneic tissue/solid organ transplantation, bone marrow transplantation, or dual umbilical cord blood transplantation.
17. Patients who, in the judgment of the principal investigator, are unlikely to comply with the trial procedures, restrictions, and requirements.
18. Patients currently enrolled in another clinical trial and receiving an investigational drugs or medical device, or those who have used any investigational drugs or device within 3 weeks prior to the first administration of the study treatment.
19. Patients who have entered the follow-up phase of a clinical trial may participate in this study only if at least 3 weeks have passed since their last use of an investigational drug or device.

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 5 years
  From randomization to time of first progression or death

SECONDARY OUTCOMES:
Overall survival | From randomization to the date of death from any cause, assessed up to 5 years
  From randomization to death.
Cancer specific survival | From date of randomization until the date of death due to ovarian cancer, assessed up to 5 years
  Cancer specific survival: From randomization to death from ovarian cancer
Adverse Event | 1 day after surgery, recovery period (3-5 weeks after surgery), up to 6 weeks after completion of chemotherapy
Health-related quality of life (EORTC-QLQ-C30) | Over the 5 year surveillance period
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
Health-related quality of life (EORTC-QLQ-OV28) | Over the 5 year surveillance period
  The EORTC QLQ-OV28 is a specified questionnaire for patients with ovarian cancer. Participant responses to the question are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized so that scores range from 0 to 100. A lower score indicates a better outcome.
Health-related quality of life (EQ-5D-5L) | Over the 5 year surveillance period
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5).
CA-125 KELIM Model | Over the 5 year surveillance period
Economic and cost evaluation | At the time of completion of 5-year surveilance period

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea